CLINICAL TRIAL: NCT04517370
Title: CO2 Laser Therapy for the Treatment of GSM in Patients With Breast Cancer A Comparative, Randomized, Controlled Trial
Brief Title: CO2 Laser Therapy for the Treatment of GSM in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 0392-18-HMO
Record Dates: First submitted 2020-08-16; First posted 2020-08-18 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Genitourinary Syndrome of Menopause
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser treatment (Active Comparator): Each patient will be treated once every 20-40 days, for a total of 3 laser treatments. In every visit during the study, patients will undergo gynecological examination and will complete questionnaires evaluating GSM symptoms, using a visual analogue scale (VAS) for each symptom (vaginal dryness, dyspareunia, discharge, itching and/or stinging, vaginal bleeding and dysuria) as well as treatment induced pain and side effects.
  Interventions: Device: Fractional/Pixel CO2 laser
- Sham treatment (Sham Comparator): Each patient will be treated once every 20-40 days, for a total of 3 Sham treatments, in a similar procedure not using an active laser energy. Patients will be assessed in a similar manner.
  Following 3 Sham-treatments patients in the placebo group will be offered the laser treatment in an open-label study .
  Interventions: Device: Fractional/Pixel CO2 laser

INTERVENTIONS:
Device: Fractional/Pixel CO2 laser — The treatment is done with a specialized vaginal applicator which allows treatment of vagina, using the Femilift fractional micro ablative CO2 laser system (Alma Lasers, Israel), according to the usual protocol (Laser mode: Pulse, Energy: 40-80 mj/pulse).
  Before treatment, 5ml of topical anesthetic ointment (10% lidocaine in Vaseline base) will be spread in the vagina and on the vestibule for 30 minutes in both groups to avoid pain from the laser, as well as to allow the comparison between the groups (patients in both groups will not experience pain and therefore will remain blinded to their allocation).

SUMMARY:
Given the need for an effective, non-hormonal treatment for Genitourinary syndrome of menopause GSM) symptoms in breast cancer survivors, the reported efficacy of fractional CO2 laser as such a treatment in retrospective studies, the study aims to evaluate the efficacy of CO2 laser for the treatment of GSM in breast cancer patients, in a prospective, randomized, blinded, placebo-controlled trial.

ELIGIBILITY:
Inclusion criteria:

1. Patients diagnosed with breast cancer
2. Menopause: spontaneous, surgical or chemotherapy induced
3. One or more GSM Symptoms: dryness, irritation, burning, pain, dyspareunia, dysuria
4. On exam, clinical findings of atrophy: thin, dry, pale vagina
5. Age>18
6. Normal Pap smear within 3 years

Exclusion criteria:

1. Menstruation
2. Chemotherapy
3. Vaginal bleeding which did not underwent evaluation
4. Concurrent treatment with topical estrogen
5. Previous vulvar, vaginal or cervical dysplasia\ cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in dryness | Follow up after 3 treatments and at 1 month, 3 months and 6 months after last treatment.
  Change in VAS before and after completion of treatment for dryness
Change in dyspareunia | Follow up after 3 treatments and at 1 month, 3 months and 6 months after last treatment.
  Change in VAS before and after completion of treatment for dyspareunia

CONTACTS AND LOCATIONS:
Overall Officials: Ahinoam Lev-Sagie, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Ahinoam Lev-Sagie, Lapid, Israel

IPD SHARING:
Plan to Share IPD: No